CLINICAL TRIAL: NCT05827718
Title: Testing Promising Behavioral Economic Interventions to Promote Enrollment Diversity in Cardiovascular Cohort Studies
Acronym: BETTER P2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: American Heart Association (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: 962643
Record Dates: First submitted 2023-03-23; First posted 2023-04-25 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: RCT #1: three-arm trial of three methods to contact patients (text v. email v. email+text) / RCT #2: two-arm trial of two sources of contact (personal clinic v. research team) / RCT #3: three-arm trial of framing methods (appeal to altruism vs. appeal to social proof vs. neither) / RCT #4: five-arm trial of incentive structure (no incentive vs. guarantee only vs. guarantee + small lottery vs. mid lottery only vs. large lottery only)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients, investigators, and outcomes assessors will all be blinded to who arm each patient is enrolled into.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- RCT #1, Arm #1: Contact Method, Text Only (Active Comparator): Potential participants in the parent trial will be randomized to receive a message via text message. This message will invite them to participate in the parent trial.
  Interventions: Behavioral: Method of Contact
- RCT #1, Arm #2: Contact Method, Email Only (Active Comparator): Potential participants in the parent trial will be randomized to receive a message via email. This message will invite them to participate in the parent trial.
  Interventions: Behavioral: Method of Contact
- RCT #1, Arm #3: Contact Method, Email+Text (Active Comparator): Potential participants in the parent trial will be randomized to receive a message via email and text message. This message will invite them to participate in the parent trial.
  Interventions: Behavioral: Method of Contact
- RCT #2, Arm #1: Source of Contact, Personal Clinic (Active Comparator): Potential participants in the parent trial will be randomized to receive a message inviting them to participate in the parent trial. The sender of the message will be the person's personal clinic.
  Interventions: Behavioral: Source of Contact
- RCT #2, Arm #2: Source of Contact, Research Team (Active Comparator): Potential participants in the parent trial will be randomized to receive a message inviting them to participate in the parent trial. The sender of the message will be the research team.
  Interventions: Behavioral: Source of Contact
- RCT #3, Arm #1: Framing Method, Appeal to Altruism (Active Comparator): Potential participants in the parent trial will be randomized to receive a message inviting them to participate in the parent trial. The message will appeal to the person's altruism, for example: "Research studies like this one often do not include enough Black individuals. If Black people are not included in research like this, then doctors have less information about how cardiovascular disease might affect them and how new treatments could be used to improve their health. Your participation in this research can help doctors better understand how to treat members of your community in the future."
  Interventions: Behavioral: Framing Method (Appeal to Altruism or Social Proof
- RCT #3, Arm #2: Framing Method, Social Proof (Active Comparator): Potential participants in the parent trial will be randomized to receive a message inviting them to participate in the parent trial. The message will include language about social proof, i.e. information about participation of individuals similar to the person being contacted. For example, the message will include language such as: "Clinical research studies and the development of effective new medications would not have been possible without the participation of thousands of people like you".
  Interventions: Behavioral: Framing Method (Appeal to Altruism or Social Proof
- RCT #3, Arm #3: Framing Method, No Appeal to Altruism, No Social Proof (No Intervention): Potential participants in the parent trial will be randomized to receive a message inviting them to participate in the parent trial. The message will include no language about appeal to altruism or social proof.
- RCT #4, Arm #1: Incentive Structure, No Incentive (No Intervention): Potential participants in the parent trial will be randomized to receive a message inviting them to participate in the parent trial. The message will have no language about incentives.
- RCT #4, Arm #2: Incentive Structure, Guarantee Only (Active Comparator): Potential participants in the parent trial will be randomized to receive a message inviting them to participate in the parent trial. The message will state that, if the person decides to participate, they will receive $25.
  Interventions: Behavioral: Incentive Structure
- RCT #4, Arm #3: Incentive Structure, Guarantee + Small Lottery (Active Comparator): Potential participants in the parent trial will be randomized to receive a message inviting them to participate in the parent trial. The message will state that, if the person decides to participate, they will receive $15 and have a 1 in 20 chance to receive $200.
  Interventions: Behavioral: Incentive Structure
- RCT #4, Arm #4: Incentive Structure, Mid Lottery Only (Active Comparator): Potential participants in the parent trial will be randomized to receive a message inviting them to participate in the parent trial. The message will state that, if the person decides to participate, they will have a 1 in 20 chance to receive $500.
  Interventions: Behavioral: Incentive Structure
- RCT #5, Arm #5: Incentive Structure, Large Lottery Only (Active Comparator): Potential participants in the parent trial will be randomized to receive a message inviting them to participate in the parent trial. The message will state that, if the person decides to participate, they will have a 1 in 100 chance to receive $2500.
  Interventions: Behavioral: Incentive Structure

INTERVENTIONS:
Behavioral: Method of Contact — Behavioral Intervention studied here is the method of contact (text vs. email vs. email+text).
  Arms: RCT #1, Arm #1: Contact Method, Text Only; RCT #1, Arm #2: Contact Method, Email Only; RCT #1, Arm #3: Contact Method, Email+Text
Behavioral: Source of Contact — Behavioral Intervention studied here is source of contact (personal clinic vs. research team)
  Arms: RCT #2, Arm #1: Source of Contact, Personal Clinic; RCT #2, Arm #2: Source of Contact, Research Team
Behavioral: Framing Method (Appeal to Altruism or Social Proof — Behavioral Intervention studied here is the framing methods "appeal to altruism" and "social proof"
  Arms: RCT #3, Arm #1: Framing Method, Appeal to Altruism; RCT #3, Arm #2: Framing Method, Social Proof
Behavioral: Incentive Structure — Behavioral Interventions studied here are guaranteed vs. lottery incentives
  Arms: RCT #4, Arm #2: Incentive Structure, Guarantee Only; RCT #4, Arm #3: Incentive Structure, Guarantee + Small Lottery; RCT #4, Arm #4: Incentive Structure, Mid Lottery Only; RCT #5, Arm #5: Incentive Structure, Large Lottery Only

SUMMARY:
Problem. Randomized clinical trials (RCTs) are the best way to determine if interventions are safe and effective. Usually only a small number of eligible patients enroll. This is because trials require people to consent to be enrolled and randomized. Black and Hispanic people are more likely to develop heart disease. They are also more likely to have risk factors for heart disease that are not controlled. Yet they are very under-represented in heart disease trials. This raises concerns about if trial results can be applied to the general population. Trial sponsors are required to enroll patients that reflect the racial and ethnic diversity of real-world people. Black and Hispanic people continue to enroll in trials at a lower rate. The goal of this study is to conduct a series of small randomized trials to test recruitment strategies to increase how many Black and Hispanic people enroll in heart disease clinical trials without diminishing trust. The investigators will test different recruitment strategies for participant enrollment in a few different areas. They will study the method of outreach, the way messages are framed, defaults, and enrollment incentives. They will run smaller recruitment strategy trials within larger parent trials (e.g. Penn Medicine Biobank cohort study). They will run a small recruitment strategy trial to test each approach and then include what they learned in the next small trial.

DETAILED DESCRIPTION:
Randomized clinical trials (RCTs) are the gold standard for determining the effectiveness and safety of drugs, medical devices, or healthcare delivery interventions. However, because RCTs require participants to consent to enrollment and randomization, typically only a minority of eligible patients enroll, raising concerns regarding the generalizability of trial results. Though Black and Hispanic individuals are disproportionately more likely to have uncontrolled risk factors for cardiovascular disease and to develop cardiovascular disease, they are substantially underrepresented in cardiovascular RCTs. In one review of 143 cardiovascular clinical trials conducted between 2008 and 2017, just 2.1% of enrollees were Black and 2.1% were Hispanic. Such low rates of enrollment have persisted despite mandates by funding and regulatory authorities that trial sponsors aim to enroll patient populations in RCTs that reflect the racial and ethnic diversity of real-world populations of patients with the disease under study. The failure of these recommendations to meaningfully increase the racial and ethnic diversity of RCT participants indicates a need for new and innovative strategies.

Behavioral economics is a scientific field of inquiry that incorporates principles from economics and psychology to better describe how individuals behave and to influence their behavior. While standard economics assumes that individuals are rational expected utility maximizers, behavioral economics recognizes that individuals' decision-making is limited by thinking capacity, available information, and time. As such, decision-making is governed by heuristics, or cognitive shortcuts. For instance, rather than trying to assess the myriad risks and benefits of participating in a research study, individuals may decide not to participate because the invitation to participate isn't from someone whose name they recognize or a perception that people like themselves do not participate. Knowledge of common heuristics can be leveraged to influence choices by modifying the context in which decisions are made, such as by changing default options or how choices are framed. Marketing studies have demonstrated the effectiveness of appeals to altruism, perceived scarcity ("This product is desirable because it is hard to get"), and social proof ("Are people like me using this product or service?") in increasing responsiveness to outreach, and these techniques can be re-purposed to increase representativeness of RCTs. Challenging social circumstances can be thought of as a "tax" on individuals' cognitive bandwidth, underscoring the opportunity to increase RCTs' racial and ethnic diversity by simplifying the enrollment process to make it easier to enroll, increasing the trustworthiness of communications, and reframing participation to make it more attractive.

The reasons for low enrollment of patients from underrepresented racial and ethnic groups in cardiovascular RCTs are multifactorial. Typically, RCTs that enroll vast majorities of patients from global regions with few Black or Hispanic patients will not enroll populations representative of U.S. demographics. Moreover, Black and Hispanic individuals are often less willing than White individuals to participate in RCTs; they are more likely to face barriers in accessing health services and to have mistrust of medical researchers, due to concerns about historic and ongoing scientific misconduct.

Newer means of communication, including patient portals, may increase or decrease representativeness depending on how they are deployed. However, few studies have systematically evaluated recruitment strategies in randomized fashion. As with any intervention, the effectiveness of different recruitment strategies is best assessed by testing different alternatives in RCTs. Accordingly, the overarching goal of this project is to conduct a series of RCTs to rigorously, systematically, and iteratively test strategies designed to increase enrollment of Black and Hispanic individuals in prospective cohort studies without diminishing trust. The investigators will embed RCTs of changes to the decision-making context, or "nudges," in the context of recruitment for prospective cohort studies because these studies' large sample size will facilitate accelerated rapid-cycle testing of multiple nudges, with results from each recruitment RCT incorporated in the next round of testing. Since the nudges are layered on top of existing cohort recruitment methods - changing only the method of outreach, message framing, or incentive structure - they are low cost, and the number of nudges that can be tested is bound primarily by the size of the cohort to be enrolled. The investigative group is uniquely positioned to conduct these studies. First, the investigators have conducted some of the only RCTs evaluating different RCT recruitment strategies. Second, they have established relationships with multiple cohort studies enrolling tens of thousands of patients with cardiovascular diseases. Third, they have extensive experience applying insights from behavioral economics to health behaviors.

The RCTs will sequentially test different strategies for participant enrollment in the following realms: method of outreach, message framing and default settings, and enrollment incentives. The primary outcome of each recruitment RCT will be the enrollment fraction of Black and Hispanic participants - the number of Black and Hispanic patients enrolled divided by the number attempted to be contacted. Because Black and Hispanic populations are heterogeneous, the investigators will also report the effect of each approach on enrollment fraction stratified according to socioeconomic status (SES), assessed using the Area Deprivation Index, a community-level SES metric. Other key secondary outcomes will include the overall enrollment fraction and the population-to-prevalence ratio, defined as the enrollment fraction of Black and Hispanic patients divided by the overall enrollment fraction. Across sequential RCTs of behaviorally-informed recruitment strategies, the investigators will accomplish the following specific aims:

Aim 1. To evaluate the effect of method of outreach on representativeness. First, patients will all receive a message via email (or traditional mail, if no email address is on file) with information about the cohort study and how to enroll and will be randomized to receive an additional message via text message or patient portal. In a subsequent RCT, potential participants will be randomized to receive this message from their personal clinic or from the research team.

Aim 2. To evaluate the effect of message framing on representativeness across two domains - appeal to altruism versus social proof versus neither. The investigators will evaluate the different framing choices in one RCT that will be embedded in an existing large cohort study.

Aim 3. To evaluate different incentive structures on representativeness. We will conduct a five-arm trial to test how incentive structure (no incentive vs. guarantee only vs. guarantee + small lottery vs. mid lottery only vs. large lottery only) affects enrollment fraction of Black and Hispanic patients.

ELIGIBILITY:
Inclusion Criteria:

* must have active medical records in site's electronic medical record system.

Exclusion Criteria:

* an electronic portal account (e.g. MyPennMedicine)
* have previously been contacted to enroll in the parent trial (e.g. Penn Medicine Biobank)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26242 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Enrollment fraction of Black + Hispanic patients | three weeks after all attempts have been made to contact is made
  The number of Black and Hispanic patients who enroll in the cohort study, divided by the total number of Black and Hispanic patients attempted to be contacted for consideration of enrollment

SECONDARY OUTCOMES:
Enrollment fraction of Black patients | three weeks after all attempts have been made to contact is made
  The number of Black patients who enroll in the cohort study, divided by the total number of Black patients attempted to be contacted for consideration of enrollment
Enrollment fraction of Hispanic patients | three weeks after all attempts have been made to contact is made
  The number of Hispanic patients who enroll in the cohort study, divided by the total number of Hispanic patients attempted to be contacted for consideration of enrollment
Enrollment fraction by Area Deprivation Index (ADI) quartile | three weeks after all attempts have been made to contact is made
  For each ADI quartile, the number of patients who enroll in the cohort study divided by the total number of patients attempted to be contacted for consideration of enrollment
Overall enrollment fraction | three weeks after all attempts have been made to contact is made
  The number of all patients who enroll in the cohort study divided by the total number of all patients attempted to be contacted for consideration of enrollment
Participation-to-prevalence ratio (PPR) for Black and Hispanic) patients | three weeks after all attempts have been made to contact is made
  The percentage of enrolled participants who identify as Black (or Hispanic) patients divided by the percentage of people who identify as Black (or Hispanic) patient in the target population.
Trust in Medical Researchers Scale | three weeks after all attempts have been made to contact is made
  Determined using the Trust in Medical Researchers Scale, a validated 4-item survey to be completed by individuals who decided to enroll in the parent trial. All four items use a 5-point Likert scale and scored accordingly (1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, 5 = strongly agree). The four items that individuals are asked to rank are: (1) Doctors who do medical research care only about what is best for each patient; (2) Doctors tell their patients everything they need to know about being in a research study; (3) Medical researchers treat people like "guinea pigs"; (4) I complete trust doctors who do medical research. The negatively-worded item (#3) is reverse-scored. So higher scores indicate more trust in medical researchers, and lower scores indicate less trust.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No